CLINICAL TRIAL: NCT07111949
Title: Investigation of the Effects of Early Skin-to-Skin Contact on Mother and Baby in Cesarean Births
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Nursing 12
Record Dates: First submitted 2025-04-17; First posted 2025-08-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-03

CONDITIONS: Skin-to-skin Contact
Keywords: skin-to-skin contact; newborn; mother; stress; cesarean delivery; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In the study, if the condition of mothers and newborns is stable immediately after the cesarean section in group 1 (SSC1), SSC will be applied as continuously as possible in the cesarean operation room, post-op care unit and ward room.
  In group 2 (SSC2), if the condition of mothers and newborns is stable after the cesarean section, SSC will be started in the post-op care unit and SSC will be continued in the ward room after the mother and baby are transferred to the maternity ward.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSC Group 1 (Operation room) (Active Comparator): Skin-to-skin contact (SSC) will be initiated in the operation room, will continue in the post-op care room, while SSC continues, the mother and baby will be transferred to the ward room, and SSC will be continued in the ward room.
  Interventions: Other: SSC Group 1 (Operation room)
- SSC Group 2 (Post-operation room) (Active Comparator): Skin-to-skin contact (SSC) will be initiated in the post-operative care unit, SSC will not be uninterrupted, SSC will be continued in the ward room.
  Interventions: Other: SSC Group 2 (Post-operation room)

INTERVENTIONS:
Other: SSC Group 1 (Operation room) — Salivary cortisol sampling from mothers, pain assessment (VAS), and measurement of physiological findings will be done at the following 3 measurement times. (1)Before transfer to the operating room (OR) (2)1 hour (h) after admission to the post-op room (PR) (3)at least 1 h after admission to the maternity ward (MW) The stress levels of the newborns will be assessed using the "Neonatal Stress Scale" at the following 4 measurement times, the heart rate and O2 saturation will be measured and recorded.
  1. At least 5 min after the initiation of SSC in the OR
  2. During the Hep-B vaccination in the PR
  3. At least 30 min after SSC after admission to the MW
  4. At least 24 h after birth in the MW, at least 30 min after SSC. The success of the newborn sucking will be assessed using the LATCH at the following 3 measurement times.
  (1) At least 5 min after the initiation of SSC in the OR (2)At least 1 h after admission to the MW, during SSC (3)At least 24 h after birth in the MW during SSC.
  Other Names: SSC1
  Arms: SSC Group 1 (Operation room)
Other: SSC Group 2 (Post-operation room) — SC sampling from mothers, pain assessment (VAS), and measurement of physiological findings will be done at the following 3 measurement times. (1)Before transfer to the OR (2)1 hour (h) after admission to the PR (3)At least 1 h after admission to the MW.
  The stress levels of newborns will be assessed using the "Neonatal Stress Scale" at the following 4 measurement times, and heart rate and oxygen saturation will be measured and recorded.
  (1)At least 5 min after birth under radiant heater in the baby care room (BCR) (2)At least 10 min after being taken to the BCR during Hep-B vaccination under radiant heater (3)At least 5 min after being admitted to the maternity ward after SSC (4)5 min after being held in the mother's arms Newborn sucking success will be assessed using LATCH at the following 3 measurement times.
  (1)At least 5 min after starting SSC in the post-op care unit (2)During SSC after being admitted to the MW (3)At least 24 h after being held in the mother's arms in the MW.
  Other Names: SSC2
  Arms: SSC Group 2 (Post-operation room)

SUMMARY:
The rate of cesarean birth continues to increase in the world and in our country. As with all surgeries, the risks of cesarean birth include the possibility of bleeding and infection, prolonged recovery time after birth, delays in initiating breastfeeding and skin-to-skin contact (SSC), and increased likelihood of complications in future pregnancies.

While many hospitals apply SSC after normal births, it is known that the number of hospitals that apply SSC in the operating room after cesarean birth is very few. Factors that prevent the initiation of SSC after cesarean birth include the effect of the current operating room culture, the physiological evaluation process of the baby after birth, the presence of procedures such as measuring body weight, aspiration, and Apgar score evaluation.

Since the mother and baby are separated after cesarean birth, the mother's initiation of breastfeeding in the first hour of life may be delayed, and the duration of exclusive breastfeeding may be shortened. The 90-minute uninterrupted skin-to-skin contact during which the baby is dried and placed directly on the mother's bare chest after birth maximizes the chance that babies are physically ready to breastfeed.

Although there are studies showing the benefits of SSC application in the operating room such as breastfeeding rates, maintaining the body temperature of the newborn, reducing maternal stress levels, and increasing oxytocin levels, a limited number of studies have been reached in the literature using SSC application guidelines developed to ensure the sustainability of SSC application in the operating room, post-op care unit, and obstetrics clinic. The first contribution of this planned study to the literature will be to standardize SSC application with SSC checklists prepared for use in the cesarean operation room, post-op care unit, and obstetrics ward based on SSC application guidelines. As a second contribution, considering the conditions of the health institution where the study will be conducted, the effects of starting SSC as early as possible and applying it in the cesarean operation room, post-op care unit, and obstetrics ward on the stress level of newborns, sucking success, and pain and salivary cortisol (stress) levels of mothers will be evaluated.

DETAILED DESCRIPTION:
The main purpose of the proposed study is to evaluate the effect of SSC initiated in different units of the hospital after cesarean delivery with spinal anesthesia on the stress level of newborns, sucking success, pain and salivary cortisol (stress) levels of mothers and physiological parameters of mothers and babies.

The secondary purpose of the study is to evaluate the satisfaction levels of mothers regarding the SSC application initiated in different units of the hospital after cesarean delivery.

Hypotheses of the Study H1: Early initiated SSC is more effective than late initiated SSC in reducing the pain level of mothers after cesarean deliveries.

H2: Early initiated SSC is more effective than late initiated SSC in reducing the salivary cortisol level of mothers after cesarean deliveries.

H3: Early initiated SSC is more effective than late initiated SSC in reducing the stress level of newborns after cesarean deliveries.

H4: Early initiated SSC is more effective than late initiated SSC on the sucking success of newborns after cesarean deliveries.

H5: Early initiation of SSC is more effective than late initiation of SSC in increasing the satisfaction level of mothers after cesarean births.

ELIGIBILITY:
Inclusion Criteria:

Mothers;

* Planning a cesarean section with spinal anesthesia
* Being between the ages of 18-45
* Having a singleton pregnancy
* Being between the gestational age of 37-40 weeks
* Not having any known health problems (diabetes, gestational diabetes, hypertension, preeclampsia, renal failure, cardiac problems, psychiatric disorders, etc.)
* Agreeing to participate in the study
* Having stable general conditions and vital signs before the skin-to-skin contact procedure
* Residing in Kütahya

Newborns (0-28 days)

* Having a gestational age between 37-40 weeks
* Having a birth weight between 2500-4500 grams
* 1-5. Apgar score ≥ 7 per minute
* No health problems, anomalies or congenital diseases
* No conditions that prevent sucking such as frenulum (tongue tie) or palate problems

Exclusion Criteria:

* Caesarean births performed with general anesthesia
* Normal births

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women with gestational age 37 and above
Enrollment: 120 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Stress levels and sucking success of newborns | From birth to the first 24 hours of life
  Newborn Stress Scale The scale items are grouped into eight subgroups using a three-point Likert scale, including facial expression, skin color, respiration, activity level, soothability, muscle tone, extremities, and posture. Each subgroup is scored on a scale of 0-2 points, with a minimum score of 0 and a maximum score of 16. As the score increases, the infant's stress level increases.
Pain and salivary cortisol (stress) levels of mothers | From before transfer to the operation room until 1 hour after transfer to the ward room after birth.
  The level of pain experienced by mothers will be assessed using a Visual Analog Scale (VAS).
  VAS is frequently used to measure subjective parameters. VAS is a 10 cm ruler where "0" represents "no pain" and '10' represents "very severe pain." The patient is instructed to mark the appropriate point on the line corresponding to the intensity of their pain. The distance from the lowest VAS level to the patient's mark is measured with a ruler in centimeters (cm) or millimeters (mm) to obtain the numerical value of the patient's pain intensity.
  Pain also causes stress. Saliva samples, a noninvasive biomarker, will be collected to determine the stress levels of mothers.

SECONDARY OUTCOMES:
Satisfaction levels o mothers regarding SSC application after cesarean delivery with spinal anesthesia | From the first SSC application until 24 hours after birth
  Mothers will be asked to rate their satisfaction with skin-to-skin contact on a scale of 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be shared by the corresponding author if requested by the journal editorship in which the study was published.